CLINICAL TRIAL: NCT06286995
Title: Postoperative Pain Assessment After Canal Preparation by Different NiTi File Systems (A Randomized Clinical Trial)
Brief Title: Postoperative Pain Assessment After Canal Preparation by Different NiTi File Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Essam Badr El-din, Bachelor, Bachelor degree in Dental Medicine and Surgery,May 2017, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6280
Record Dates: First submitted 2024-02-24; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Pain; Inflammation
Keywords: Post operative pain; Substance P; Apical periodontitis; Trunatomy file; Edgeendo x7 file
MeSH Terms: conditions — Pain, Postoperative; Inflammation; Periapical Periodontitis | interventions — Root Canal Therapy

STUDY DESIGN:
Intervention Model Description: This study was designed to be randomized,single- blinded, single-center clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: A) Sequence generation: was done using random sequence number generated by computer software B) Allocation concealment Mechanism:folded,numbered papers were placed in tightly sealed envelopes containing patients' coding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunatomy file group (Active Comparator): Using trunatomy file for chemomechanical preparation for root canal of mandibular premolars
  Interventions: Procedure: Chemomechanical preparation for root canals
- Edgeendo x7 file group (Active Comparator): Using edgeendo x7 file for chemomechanical preparation for root canal of mandibular premolars
  Interventions: Procedure: Chemomechanical preparation for root canals

INTERVENTIONS:
Procedure: Chemomechanical preparation for root canals — After working length determination ,root canal preparation was made by two different NiTi File systems to both group ( the first group using Trunatomy file and the second one using edgeendo x7 file) and assessment of pain was made preoperatively and postoperatively and also apical fluid samples
  Other Names: Root canal treatment

SUMMARY:
The participants were divided into two groups : group one ( Trunatomy file group)(n=10) was mechanically prepared the canals by Trunatomy file and group two ( Edgeendo x7 file group) ( n=10) was prepared the canals by Edgeendo x7 file, the participants were assessed pain preoperatively and postoperatively by Visual Analog Scale(VAS)

DETAILED DESCRIPTION:
Patients : 20 patients with symptomatic apical periodontitis related to mandibular premolars were selected.after proper anathesia, Access cavity was ppreformed.The working length measured using apex locator.chemomechanical preparation was done .for trunatomy file group ,using file sequence according to manufacture's instructions until medium one .for edgeendo group ,using file sequence also according to manufacture's instructions until file size 35 taper4.Apical fluid samples was collected by paper point from the both preoperatively and before obturation and also pain was assessed pre and post opertively.finally,the root canal were filled by gutta-percha and resin based sealer.the access cavity was restored by glass ionomer restoration.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnoses of apical periodontitis related to single-rooted mandibular premolars
* no evidence of excessive mobility

Exclusion Criteria:

* presence of any systemic disease or allergic reaction
* Incompletely formed root
* Previously Endodontically treated teeth

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Level of post operative pain using 10-cm visual analogue scale ( VAS) | After 6 hours,24 hours, 48 hours and finally 72 hours
  10-cm visual analogue scale (VAS) questionnaire.each patient reported their level of pain as follow: 0 no pain,1-3 mild pain,4-6 moderate pain,7-9 severe pain and 10 the worst pain

SECONDARY OUTCOMES:
Level of inflammatory mediators substance P in apical fluid samples | Preoperatively ( after working length determination) and before obturation after 3days
  Sample were obtained by paper point size 25passing 2mm beyond the apex where they were soaked in the periapical interstitial fluid for 1minute .four mm from tip of paper point we're cut and dropped into 1,5ml Eppendorf tubes ( Swanscombe,UK) with 1ml of phosphate buffered saline,then restored at -80 to be measured by ELISA test

CONTACTS AND LOCATIONS:
Overall Officials: Maram F Obeid, Professor, Study Director — Faculty of dentistry, Ain shams university
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Detailed statistical analysis plan
Supporting Information: SAP
Time Frame: 2025, available for a year
Access Criteria: Review the purpose of request
URL: http://asmj.journal.ekb.eg

REFERENCES:
- [Background] Caviedes-Bucheli J, Azuero-Holguin MM, Gutierrez-Sanchez L, Higuerey-Bermudez F, Pereira-Nava V, Lombana N, Munoz HR. The effect of three different rotary instrumentation systems on substance P and calcitonin gene-related peptide expression in human periodontal ligament. J Endod. 2010 Dec;36(12):1938-42. doi: 10.1016/j.joen.2010.08.043. Epub 2010 Oct 15. PMID 21092809
- [Background] Valliappan CT, Rahul B, Gabriel EM, Sherwood IA, Gutmann JL, Amaechi BT, Burhanuddin Mohammed OF. Evaluation of postoperative pain with new heat-treated rotary and reciprocating nickel-titanium files: A randomized controlled clinical trial. J Conserv Dent. 2023 Mar-Apr;26(2):170-175. doi: 10.4103/jcd.jcd_566_22. Epub 2023 Mar 16. PMID 37205884
- See also: Worked on inflammatory mediators in similar matter — http://dsu.journals.ekb.eg/article_192084.html